CLINICAL TRIAL: NCT06763887
Title: Evaluation of Immunogenicity of COVID-19 Vaccine in Chinese Population
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20232379-C-1
Record Dates: First submitted 2024-11-21; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Observation
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No intervention

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and immune protection of COVID-19, especially the recently prevalent strains, against the background of current immunization in Chinese population

ELIGIBILITY:
Inclusion Criteria:

1. He was infected with COVID-19 from November to December 2022;
2. Have not been infected with COVID-19 (the subject said that he was not infected and signed the informed consent form);
3. Those who agree and sign the informed consent form.

Exclusion Criteria:

1. Missing or incomplete questionnaires that affect research results;
2. Individuals with combined dysfunction of important organs such as the heart, liver, and lungs;
3. Mental and behavioral abnormalities;
4. Intellectual disability;
5. Under 18 years old or over 75 years old;
6. Low understanding and communication skills.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People infected with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
PBMC | About two and a half years
  When conducting blood sample analysis, we focus on separating and evaluating in detail the composition and counting of peripheral blood mononuclear cell (PBMC). This process involves identifying and quantifying various types of mononuclear cells in the sample, such as lymphocytes, monocytes, etc. These cells are crucial for understanding an individual's immune status. Through precise separation techniques and advanced cell analysis methods, we are able to obtain accurate and detailed reports on the classification and quantity of mononuclear cells.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Air Force Military Medical University, Xi'an, Shaanxi, China